CLINICAL TRIAL: NCT01262989
Title: Randomized, Two-period, Cross-over, Bioequivalence Study on Tamsulosin Hydrochloride 0,4 mg Prolonged Release Hard Gelatin Capsule Versus SECOTEX® (Tamsulosin Hydrochloride) 0,4 mg Prolonged Release Hard Gelatin Capsule (Boehringer Ingelheim) in Healthy Male Volunteers Under Fasting Conditions.
Brief Title: SECOTEX® (Tamsulosin Hydrochloride) Bioequivalence Study Brazil - Fast Admin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 114071
Record Dates: First submitted 2010-09-03; First posted 2010-12-20 (Estimated); Results first posted 2011-03-31 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Prostatic Hyperplasia
Keywords: Bioequivalence; Tamsulosin; Healthy volunteers; Fast conditions
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tamsulosin Reference (Active Comparator): Reference drug administration followed by Test drug administration
  Interventions: Drug: Test formulation; Drug: Reference formulation
- tamsulosin Test (Active Comparator): Test drug administration followed by Reference drug administration
  Interventions: Drug: Test formulation; Drug: Reference formulation

INTERVENTIONS:
Drug: Test formulation — tamsulosin hydrochloride 0,4 mg (Synthon BV)
Drug: Reference formulation — tamsulosin 0,4 mg (Boehringer Ingelheim)

SUMMARY:
It will be an open-label, randomized, laboratory-blind, crossover study with 02 treatments, 02 sequences, and 02 periods, in which the healthy male volunteers under fasting conditions receive, in each period, the test formulation or the reference formulation

DETAILED DESCRIPTION:
TITLE: Randomized, two-period, cross-over, bioequivalence study on tamsulosin hydrochloride 0,4 mg prolonged release hard gelatin capsule (Synthon BV, The Netherlands) versus SECOTEX® (tamsulosin hydrochloride) 0,4 mg prolonged release hard gelatin capsule (Boehringer Ingelheim do Brasil Química e Farmacêutica Ltda) in healthy male volunteers under fasting conditions.

It will be an open-label, randomized, laboratory-blind, crossover study with 02 treatments, 02 sequences, and 02 periods, in which the healthy male volunteers under fasting conditions receive, in each period, the test formulation or the reference formulation.

The treatment's sequence attributed to each volunteer on the study period is determined by a randomization list, which is generated by PROC PLAN from SAS version 9.1.3 system.

The formulations will be administered as a single oral dose followed by blood collections between, at least, 3 to 5 half-lives. The treatment's periods may obey a minimum interval of 7 half lives between them (period for drug's whole elimination by the organism).

ELIGIBILITY:
EXCLUSION CRITERIA:

* Known hypersensitivity to the study drug (tamsulosin hydrochloride) or to compounds chemically related
* History or presence of hepatic or gastrointestinal illnesses, or other condition that interferes over the drug's absorption, distribution, excretion or metabolism
* History of hepatic, renal, pulmonary, gastrointestinal, epileptic, hematologic or psychiatric illness
* Hypotension or hypertension of any etiologic that needs pharmacologic treatment
* Volunteer has history or had myocardial infarction, angina and/or heart insufficiency
* Non-recommended electrocardiographic findings, according investigator criteria
* The results of the laboratory exams are out of the values considered as normal according this protocol's rules, unless that they are considered as clinically irrelevant by the investigator
* Volunteer is a smoker
* The volunteer ingests more than 5 cups of coffee or tea a day
* History of alcohol or drugs abuse
* History of serious adverse reactions or hypersensitivity to any drug
* Use of any regular drug within the 02 weeks that preceded study's initiation or treatment within the 03 previous months, that preceded study's initiation, with any drug that presents toxic, or consumed inductive drugs and/or enzymatic inhibitors (CYP450 - hepatic), within the 04 weeks that preceded the study's initiation
* Hospitalization for any reason within 08 weeks of beginning of the study's first period of treatment and the post study assessment date
* Participation in any experimental study or ingested any experimental drug within the 06 previous months
* Donation or lost of 450mL or more of blood within the 03 previous months
* Volunteer consumed alcohol in 48 hours prior to the admission to the study or consumed foods or beverages that contain grapefruit until 07 days previous to each study period

INCLUSION CRITERIA:

* Male
* Age between 18 and 50 years
* Body mass index ≥ 19 and ≤28,5
* Good health conditions or without significant illness, by judgment of a legally qualified professional, according the rules defined in Protocol, and according the following evaluations: clinical history, pressure and pulse measures, physical and psychological exam, ECG, and additional laboratory exams
* Capable to understand the study's nature and aim, including the risks and adverse effects and with intention to cooperate with the researcher and to act in compliance with the requirements of the whole assay; this will be confirmed by the Informed Consent's signature.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01-04 (Actual); Primary Completion 2010-01-26 (Actual); Study Completion 2010-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Campinas, São Paulo, Brazil

REFERENCES:
- See also: Results for study 114071 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114071?search=study&search_terms=114071#rs

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product in Period 1; Reference Product in Period 2: Test product: tamsulosin hydrochloride 0.4 milligrams (mg) prolonged release hard gelatin capsule, once a day, in Period 1 (duration of 3 days); followed by a 7-day washout period during which no medication was administered; followed by reference product: SECOTEX (tamsulosin hydrochloride) 0.4 mg prolonged release hard gelatin capsule, once a day, in Period 2 (duration of 3 days)
- Reference Product in Period 1; Test Product in Period 2: Reference product: SECOTEX (tamsulosin hydrochloride) 0.4 mg prolonged release hard gelatin capsule, once a day, in Period 1 (duration of 3 days); followed by a 7-day washout period during which no medication was administered; followed by test product: tamsulosin hydrochloride 0.4 mg prolonged release hard gelatin capsule, once a day, in Period 2 (duration of 3 days)
Period: Period 1
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 20 | 20
Completed | 19 | 17
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Intercurrent disease | 0 | 1
Not completed — Positive answer for exclusion criteria | 0 | 1
Period: 7-Day Washout Period
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 19 | 17
Completed | 19 | 16
Not Completed | 0 | 1
Not completed — Intercurrent disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants Receiving Both Test Product and Reference Product: Participants receiving either test product: tamsulosin hydrochloride 0.4 mg prolonged release hard gelatin capsule, once a day, in Period 1 (duration of 3 days); followed by reference product: SECOTEX (tamsulosin hydrochloride) 0.4 mg prolonged release hard gelatin capsule, once a day, in Period 2 (duration of 3 days) or reference product in Period 1 and test product in Period 2
Arm/Group | Participants Receiving Both Test Product and Reference Product
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.65 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 34
  Mulatto | 5
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC from time 0 (prior to administration of medication) to time t (the time of the last quantifiable concentration) was calculated using the trapezoidal method. This method consists of the sum of the trapezoids' areas, determined by the collection times and their concentrations. The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. ng, nanograms; ml, milliliter.
Time Frame: Days 1 to 3 (Period 1) and Days 9 to 11 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng per hour per ml (ng/h/ml)
Groups:
- Test Product: Test product tamsulosin hydrochloride 0.4 milligrams (mg) prolonged released hard gelatin capsule, once a day, in both periods (duration of 3 days in each period)
- Reference Product: Reference product SECOTEX (tamsulosin hydrochloride) 0.4 mg prolonged release hard gelatin capsule, once a day, in both periods (duration of 3 days in each period)
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 35 | 35
ng per hour per ml (ng/h/ml) | 237.35 (115.56) | 226.74 (103.34)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — This is a bioequivalence study performed to support the register of tamsulosin hydrochloride, produced by Synthon BV, as a branded generic, to be marketed by GlaxoSmithKline Brasil Ltda., according to the requirements of the Brazilian Regulatory Agency - National Agency of Sanitary Surveillance (ANVISA); Ratio T formulation/R formulation = 102.95, 90% CI [97.17 to 109.07] — The ratios between the geometric means of the test (T) and reference (R) formulations was calculated

2. Primary Outcome: AUC0-infinity
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC from time 0 (prior to administration of medication) to infinity (the time of complete elimination of the drug) was calculated using the trapezoidal method. This method consists of the sum of the trapezoids' areas, determined by the collection times and their concentrations. The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption.
Time Frame: Days 1 to 3 (Period 1) and Days 9 to 11 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng/h/ml
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 35 | 35
ng/h/ml | 244.00 (119.49) | 233.34 (107.11)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 102.79, 90% CI [96.99 to 108.93] — The ratios between the geometric means of the test (T) and reference (R) formulations was calculated

3. Primary Outcome: Cmax
Description: Cmax is defined as the maximum or "peak" concentration of a drug observed after its administration. Cmax is one of the parameters of particular use in estimating bioavailability of drugs, by measuring the total amount of drug absorbed.
Time Frame: Days 1 to 3 (Period 1) and Days 9 to 11 (Period 2)
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 35 | 35
ng/ml | 20.27 (9.54) | 20.80 (7.86)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 94.47, 90% CI [87.59 to 101.90] — The ratios between the geometric means of the test (T) and reference (R) formulations was calculated

ADVERSE EVENTS:
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product in Period 1; Reference Product in Period 2 (N=20) | Reference Product in Period 1; Test Product in Period 2 (N=20)
Fever (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Serum glutamic-pyruvic increased (Investigations) | 0 | 4
Gamma glutamyl transferase increased (Investigations) | 0 | 4
Serum glutamic-oxaloacetic increased (Investigations) | 0 | 1
Serum cholesterol increased (Investigations) | 0 | 1
Serum urea increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Lumbago (Musculoskeletal and connective tissue disorders) | 1 | 0
Extremities burning sensation (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 7 | 2
Throat pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.